CLINICAL TRIAL: NCT06469619
Title: The Effect of Music Listening in Rehabilitation of Subacute Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maria Sariola (Other)
Responsible Party: Sponsor-Investigator, Maria Sariola, Neurologist, Tampere University Hospital
Organization: Tampere University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R24013
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Physiotherapists, occupational therapists and speech therapists who are responsible for rehabilitation and perform the testing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Standard care and rehabilitation.
- Music group (Experimental): Standard care and rehabilitation and music listening one hour a day during 4 weeks.
  Interventions: Behavioral: Music listening

INTERVENTIONS:
Behavioral: Music listening — Listening to music of one's choice one hour daily.
  Arms: Music group

SUMMARY:
Music listening has many positive effects on the brain. This study aims to find out if people with stroke get better results with their rehabilitation if they listen to music during their passive hours. The study is a randomized controlled trial with people who are at a rehabilitation center care after stroke at Tampere University Hospital. The control group gets standard rehabilitation. Music group gets standard rehabilitation and in addition they listen to music one hour a day during four weeks. Physiotherapists, occupational therapists and speech therapists test how well the participant's walking, use of hand and speech improve. The main goal is to find out if the improvement is better with music listening. The study also monitors effects of music listening on mood in rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* hemispheric stroke (ischemic or intracerebral hemorrhage) during last 4 weeks OR spinal cord injury in last 6 months, causing a need of intensive rehabilitation

Exclusion Criteria:

* severe hearing loss preventing music listening
* previous condition of neurological disease of dementia that significantly affects daily functions
* active drug use or acute psychiatric condition
* unable to understand given information and give consent to participate
* for spinal cord injury patients: acute traumatic brain injury or stroke

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in lower extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  Functional Ambulation Classification
Change in lower extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  Berg balance scale
Change in lower extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  10 m walking test
Change in lower extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  Timed Up and Go
Change in upper extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  Box and Block
Change in upper extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  9-hole Peg Test
Change in upper extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  Grip strength
Change in upper extremity function | At time point 0 and 4-5 weeks later (Before and after intervention)
  Arm abduction (scale 1-3, 1 = normal, 2 = able to lift between horizontal plane but with at least 30 degrees deficiency, 3 = unable to lift above horizontal plane)
Change in speech | At time point 0 and 4-5 weeks later (Before and after intervention)
  Boston Naming Test
Change in speech | At time point 0 and 4-5 weeks later (Before and after intervention)
  Western Aphasia Battery
Change in speech | At time point 0 and 4-5 weeks later (Before and after intervention)
  Token
Change in speech | At time point 0 and 4-5 weeks later (Before and after intervention)
  Story based on a nine-frame cartoon (standardized point scale)
Mood | At time point 0 and 4-5 weeks later (Before and after intervention)
  Visual Analogue Mood Scale
Mood | At time point 0 and 4-5 weeks later (Before and after intervention)
  Beck Depression Inventory
Mood | At time point 0 and 4-5 weeks later (Before and after intervention)
  Generalized Anxiety Disorder-7
Daily functions | At time point 0 and 4-5 weeks later (Before and after intervention)
  Rivermead Motor Assessment Gross function
Daily functions | At time point 0 and 4-5 weeks later (Before and after intervention)
  Functional Status Questionnaire (FSQfin)

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Palmio, Principal Investigator — The Wellbeing Services County of Pirkanmaa, Tampere University

IPD SHARING:
Plan to Share IPD: No